CLINICAL TRIAL: NCT07122180
Title: Post-Market Clinical Follow-Up of the CT3 Series Continuous Glucose Monitoring System: A 14-Day Observational Study Assessing Accuracy, Safety, and Glucose Control in Patients With Type 1 and Type 2 Diabetes Mellitus
Status: Enrolling by invitation | Type: Observational
Sponsor: MDCECRO LLC (Network)
Responsible Party: Sponsor
Other Study IDs: Yuw-CGM-20250306
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CT3 Series Continuous Glucose Monitoring System: — The CT3 Series CGM System is a real-time, continuous glucose monitoring device indicated for the management of diabetes in adults (age≥18 years). Interpretation of the CT3 Series CGM System results should be based on the glucose trends and several sequential readings over time. The CT3 Series CGM System also aids in the detection of episodes of hyperglycaemia and hypoglycaemia. It is intended for single-patient use. It is intended to replace fingerstick blood glucose testing for diabetes treatment decisions unless otherwise indicated

SUMMARY:
Post market Clinical follow-up of the CT3 Series Continuous Glucose Monitoring System: A 14-Day Observational Study Assessing Accuracy, Safety, and Glucose Control in patients with Type 1 and Type 2 Diabetes Mellitus

DETAILED DESCRIPTION:
To re-assess the benefits of CT3 series CGM and the risks of skin abnormalities, hypoglycaemia, hyperglycaemia so as to improve CT3 series CGM continuously.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients diagnosed with type 1 or 2 diabetes mellitus. 2.People aged 18 years or older, regardless of gender. 3.Those who sign informed consent to participate in this study voluntarily. 4.The patient had good compliance and could complete this whole clinical investigation.

Exclusion Criteria:

* 1.Those who have broken, scarred, red, swollen, or infected skin on the upper arms or abdomen.

  2.Those who are allergic to alcohol disinfectants or medical adhesive tapes. 3.Those who have hematologic diseases that affect coagulation function or have been diagnosed with a bleeding tendency.

  4.Those who have anemia or abnormal hematocrit. 5.Pregnant and lactating women. 6.Psychiatric abnormalities, cognitive and communication disorders, or highly stressed and uncooperative.

  7.Those with subcutaneous edema at the wearing site. 8. Those who plan to undergo magnetic resonance imaging (MRI), computed tomography (CT), or X-ray examination within 14 days of wearing.

  9. Those who have participated in clinical trials of drugs or devices within 1 month.

  10.Those who are considered by the investigator to be inappropriate to participate in this PMCF study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with type 1 or 2 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2025-09-17 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
This PMCF study (Version V2.0) uses a strong evaluation plan, with methods and timing carefully matched to the study's rules. It includes 72 patients | 14 days
  The Continuous Glucose Monitoring (CGM) is done for 14 days for each person. During this time, glucose readings are collected every three minutes in real-time Self-Monitoring of Blood Glucose (SMBG) involves using fingerstick tests to check glucose levels.
  Important measurements-like Time in Range (TIR), Time Above Range (TAR), Time Below Range (TBR), and error grid analysis-are taken at specific times, including at the beginning and on certain follow-up days.
  These timings help collect key data to check how well the device works in the short term and how it affects glucose control over the full monitoring period.

CONTACTS AND LOCATIONS:
Locations (1):
- Paula Stradiņa klīniskā universitātes slimnīca, Riga, Rīga, Latvia

IPD SHARING:
Plan to Share IPD: Undecided